CLINICAL TRIAL: NCT07379983
Title: Evaluating the Effectiveness of Print Based Environmental Health Intervention Education Among School Going Adolescents of Karachi, A Quasi Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Hina Sharif, Senior Lecturer, Bahria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00008
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Environmental Health; Adolescent Health; Green Spaces; Plantation; Waste Management; Educational Intervention; Water-Borne Infectious Disease; Safe Water
MeSH Terms: conditions — Waterborne Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effectiveness of knowledge on environmental health, through Poster (Experimental)
  Interventions: Behavioral: Educational Intervention either from Poster or Infographic pamphlet
- effectiveness of knowledge on environmental health, through Infographic pamphlet (Experimental)
  Interventions: Behavioral: Educational Intervention either from Poster or Infographic pamphlet

INTERVENTIONS:
Behavioral: Educational Intervention either from Poster or Infographic pamphlet — Age-appropriate sessions on climate science, health impacts (heat stress, vector-borne diseases, air pollution), mindful use of water, proper waste management and local relevance (e.g., Karachi's heatwaves, dengue outbreaks)

SUMMARY:
This study investigates the impact of school-based educational interventions on adolescents' knowledge and practices related to environmental health in Karachi, Pakistan. The methodology opted for this research is quasi experiment with three months intervention period. The research will begin with a baseline survey to assess adolescents' understanding of environmental health, green spaces, waste management, and associated health impacts. Schools are then engaged in creating and maintaining green spaces and adopting waste management practices. Two intervention arms are implemented: Arm 1 receives educational content through posters, while Arm 2 receives pamphlets. In March, schools are revisited to evaluate the maintenance of cleanliness and green spaces. Finally, in April, a post-intervention survey will be conducted to measure changes in knowledge and eco-friendly practices. The study aims to determine the effectiveness of posters versus pamphlets in enhancing knowledge and sustaining environmental practices among adolescents, thereby contributing to evidence-based strategies for promoting environmental health education in urban school settings.

ELIGIBILITY:
Inclusion Criteria:

* The study will target only one mode of education in Karachi, i.e., the matriculation system, including both public and private schools to cover a broad segment of the adolescent student population.
* Schools registered with the Board of Secondary Education Karachi (BSEK) will be included, ensuring that students from both sectors will follow the same curriculum.
* Schools must have at least 30 students in each class from 6th to 10th grade, so that each class can serve as a stratum.
* Only schools that provide permission to conduct the study within their premises will be enrolled.
* Only students who provide assent and whose parents provide consent will be included

Exclusion Criteria:

* Any participant who plans to leave their school during the study period.
* Any participant who is not present during any round of the study, i.e., before and after the intervention.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Increased Knowledge about environmental Health | 3 months
  High Environmental & Health Awareness (28-36 points)
  Strong knowledge
  Excellent awareness of pollution, climate issues, and disease linkages
  Likely to engage in positive environmental behaviour
  Moderate Awareness (18-27 points)
  Good understanding but with some gaps
  Needs moderate reinforcement through school/community programs
  Low Awareness (0-17 points)
  Limited understanding
  Requires structured awareness sessions and visual learning tools

SECONDARY OUTCOMES:
Waterborne and Airborne Disease Knowledge | 3 months
  High Environmental & Health Awareness (28-36 points)
  Strong knowledge
  Excellent awareness of pollution, climate issues, and disease linkages
  Likely to engage in positive environmental behaviour
  Moderate Awareness (18-27 points)
  Good understanding but with some gaps
  Needs moderate reinforcement through school/community programs
  Low Awareness (0-17 points)
  Limited understanding
  Requires structured awareness sessions and visual learning tools

IPD SHARING:
Plan to Share IPD: No